CLINICAL TRIAL: NCT06277999
Title: An Observational Study in Adults With Clostridioides Difficile Infection to Determine the Feasibility and Logistics of Biospecimen Collection, Transportation and Testing at Select US Study Sites
Brief Title: C.Difficile Observational Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8820C00001
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Clostridium Infections
Keywords: Clostridiodes difficile infection, C difficile
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool, serum samples

GROUPS / COHORTS (2):
- Monitoring Cohort: Monitoring cohort will enroll a targeted minimum of 20 and a maximum of 100 participants ≥ 18 years of age who have been recently diagnosed with CDI by a licensed HCP and are receiving SOC antibiotic treatment, with treatment starting ≤ 5 days before study enrollment. Participants will be recruited from hospitals which perform C difficile laboratory diagnostic testing. Recruitment will occur over a 6-month period. Participants will be followed through Day 42, with a screening period from Day -5 to Day 1
- Discard Stool Cohort: The Discard Stool cohort will include stool specimens from up to 200 participants, ≥ 18 years of age, who have been recently diagnosed with CDI by a licensed HCP within the past 7 days. Participants in this cohort will be screened at the study site to confirm eligibility. Following the screening period, there will be no additional study activities for the participant to complete.

SUMMARY:
D8820C00001 is an exploratory, non-interventional, unblinded, observational study evaluating the acceptability, feasibility and performance of methods to collect, transport and test biospecimens in participants ≥ 18 years of age with an active CDI. Participants will also be monitored for recurring episodes of diarrhea and will need to complete validated PROs and study evaluation questionnaires

DETAILED DESCRIPTION:
The premise of D8820C00001 study is to monitor participants for recurring episodes of diarrhea and evaluate acceptability and feasibility of the use of the digital tools and patient outcome measures. The aim will be to enroll two cohorts of patients; the first will be the Monitoring cohort, enrolling a targeted minimum of 20 and a maximum of 100 participants who will be followed through Day 42, with a screening period from start of standard of care treatment to Day 1 (see Section 2.1.1). The second will be the Discard Stool cohort, enrolling up to 200 participants, who will not be followed during the study but who will provide consent for the use of any discarded stool specimens that will not be used for additional laboratory diagnostic testing .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years of age at the time of signing the informed consent
2. Participants in the Monitoring and Discard Stool cohorts with an active treated CDI, defined as meeting all of the following:

   * Prior to or at diagnosis of C. difficile, either diarrhea, defined as ≥ 3 unformed stools in a 24 hour period, with the stool being measured as Types 5, 6, 7 on the Bristol Stool Scale or evidence of megacolon, or severe ileus.
   * A positive local stool test results for toxigenic C difficile collected before entry to the study or evidence of pseudomembranes demonstrated by endoscopy or histopathology.

   For the Monitoring Cohort - positive test result immediately prior to start of or during SOC treatment.

   For the Discard Stool Cohort - no more than 7 days prior to entry to the study.
   * Stool test positive for only GDH or PCR and negative for toxin, provided there is observed clinical improvement noted by the Investigator within 5 days of start of SOC treatment, characterized by a reduction in diarrhea , in the the judgement of the Investigator
   * Receiving SOC therapy for the treatment of CDI at the time of enrollment.
3. Able to complete all study assessments, and to understand and comply with study requirements/procedures (if applicable, with assistance by caregiver, surrogate, or legally authorized representative, or equivalent representative as locally defined) based on the assessment of the PI
4. Able to complete the Follow-up period through Day 42 based on the assessment of the PI.
5. If able, signed and dated written informed consent prior to any study specific procedures, including screening evaluations for participants who consent to participate in the Monitoring cohort. Ensure that participants who are considered by the Investigator clinically unable to consent at screening and who are entered into the study by the consent of a legally acceptable representative show evidence of assent, as applicable in accordance with local regulations.
6. Signed and dated written information consent prior to collection and testing of stool samples for participants in the Discard Stool cohort

Exclusion Criteria:

1. Employees of AstraZeneca, clinical study site, or any other individuals directly involved with the conduct of the study, or immediate family members of such individuals. Employees of the clinical site or immediate families of these individuals not directly involved in the clinical study will be permitted to participate.
2. Deprived of freedom by an administrative or court order, or in emergency setting, or hospitalized involuntarily
3. Absence of suitable venous access for serum sampling

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥ 18 Years of Age (Adult, Older Adult )
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Number of participants that completed key study activities according to protocol | from Day 1 to Day 42
  Evaluation of the overall and individual completion rate of procedures and logistics involved in key study activities defined as:
  * Stool sample collection, transport, and processing.
  * Serum collection.
  * Identification of suspected rCDI using the participant monitoring strategy
  * Cdiff32, CDI-DaySyms and PGI-S PRO questionnaire completion rate during the SOC treatment period.

SECONDARY OUTCOMES:
Time intervals across stool sample collection logistics | from Day 1 to Day 42
  All stools counted regardless of multiple stools per participant:
  * selected percentiles of empirical distribution of time taken for samples to be collected by courier for transport to central lab (split by geography, site, or home)
  * selected percentiles of empirical distribution of time taken of testing procedure or components thereof
Participant Experience and site staff evaluation questionnaires | from Day 1 to Day 42
  Review of Participant Experience and site staff evaluation questionnaires for qualitative and quantitative feedback on factors which affect completion of study activities, including participant acceptability of study activities
Gather information to assess logistics, resourcing and performance of different toxin detection assays (eg. EIA, PCR, CCNA) | from Day 1 to Day 42
  Number of samples completed in accordance to study protocol, time to complete testing, number of samples tested with stability window

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, Sacramento, California
  - Research Site, Hamden, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Charleston, South Carolina
  - Research Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8820C00001&attachmentIdentifier=e88473c0-97cd-4697-a5f6-cc0157300d69&fileName=D8820C00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=